CLINICAL TRIAL: NCT04099849
Title: Absorption of Zinc From Mixed Diets Containing Conventional Bangladeshi Rice, Zinc-biofortified Bangladeshi Rice, or Conventional Bangladeshi Rice With Added Zinc Among Young Children From a Peri-urban Community
Brief Title: Zinc Absorption From Zinc Biofortified Rice in Bangladeshi Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PR-13008
Record Dates: First submitted 2019-09-20; First posted 2019-09-23 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-01

CONDITIONS: Malnourished Children
Keywords: Rice; biofortification,; Bangladeshi children; zinc

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Diet-ZnBfR zinc biofortified rice-based diet
  Diet- CR conventional rice-based diet
  Interventions: Dietary Supplement: Diet-ZnBfR: Zinc biofortified rice-based diet; Dietary Supplement: Diet- CR: Conventional rice-based diet
- Group B (Experimental): Diet-ZnBfR zinc biofortified rice-based diet
  CR + Zn conventional rice-based diet plus zinc fortificant (Diet-CR+Z).
  Interventions: Dietary Supplement: Diet-ZnBfR: Zinc biofortified rice-based diet; Dietary Supplement: CR + Zn: Conventional rice-based diet plus zinc fortificant (Diet-CR+Z).

INTERVENTIONS:
Dietary Supplement: Diet-ZnBfR: Zinc biofortified rice-based diet — Diet-ZnBfR: Zinc biofortified rice-based diet
Dietary Supplement: Diet- CR: Conventional rice-based diet — Diet- CR: Conventional rice-based diet
  Arms: Group A
Dietary Supplement: CR + Zn: Conventional rice-based diet plus zinc fortificant (Diet-CR+Z). — CR + Zn: Conventional rice-based diet plus zinc fortificant (Diet-CR+Z).
  Arms: Group B

SUMMARY:
It is well documented that zinc supplementation to low-income population results in the reduced incidence of childhood diarrhoea and pneumonia, and improves growth of stunted children. In Bangladesh, the risk of zinc deficiency is considered to be high and children could benefit greatly by improving their zinc intakes on a daily basis. Zinc supplementation at a national scale would be a formidable task. There is a need to find an alternative. It might be sustainable to improve intake of zinc through fortified staples, e.g. rice with increased amounts of zinc; in fact such biofortified rice has been developed through conventional breeding, which is designed to contain an amount of zinc that could meet at least 40% of the daily requirement.

In the first round of the previously approved and completed studies, total absorbed zinc (TAZ) did not differ when diets containing zinc biofortified rice (ZnBfR) or conventional rice (CR) were compared. Thus, the current study is planned to repeat using a new variety of (ZnBfR) that is expected to have higher zinc content than the variety previously studied. Initially, a pilot study will be conducted in 4 participants using a modified isotope administration protocol such that the oral tracers will be given on two days each at half the original dose each day so as to provide a lower proportion of the total daily zinc intake as tracer solution.

Hypotheses:

1. Young children will have greater total absorbed zinc (TAZ) when they consume mixed diets containing ZnBfR than when they consume the same diets containing CR.
2. TAZ will not differ in children who receive the ZnBfR-containing diet or the same diet containing CR plus sufficient additional zinc to match the zinc content of the ZnBfR diet.

Objectives:

1. To measure the amount of zinc absorbed from ZnBfR compared with the amount absorbed from CR and from CR fortified with added zinc, using the triple stable isotope tracer ratio technique in young children.
2. To assess the intestinal function of the children, using a sugar permeability test (lactulose:mannitol test).
3. (Pilot study) To verify that the modified tracer dose will provide adequate signal for assessing zinc absorption.

Methods:

To assess the potentials for biofortified rice in providing a good, bioavailable source of additional zinc, it is proposed here to measure zinc absorption from rice-based meals among Bangladeshi preschool children. The amount of zinc absorbed from ZnBfR compared to that absorbed from a conventional Bangladeshi rice (Diet-CR) (control) will be measured. Zinc absorbed from ZnBfR with that from zinc-fortified conventional rice (Diet-CR+Z) will also be compared. The study will be a cross-over, randomized, controlled clinical study. Initially, a pilot study will be conducted with a modified dose of zinc stable isotope among 4 children aged 36-59 months of either sex from a peri-urban community in Dhaka. Later on, 44 children aged 36-59 months of either sex will be recruited from the same community as mentioned before, and they will be individually randomized, in equal numbers, to one of the two comparison groups, A and B. During an initial one-day acclimatization period, the study children will receive the conventional rice based diet three times a day, to confirm that they will accept the study diets and adhere to the study procedures. On study days 2 and 4, in comparison group A, the study subjects will receive either the Diet-ZnBfR or Diet-CR based on the random assignments, and they will receive Diet-CR or Diet ZnBfR, respectively, on days 3 and 5 (i.e., the diet not received on days 2 and 4), Likewise, in comparison group B, the study subjects will receive either Diet-ZnBfR or Diet-CR+Z on days 2 and 4 based on the random assignments, and they will receive Diet-CR+Z or the Diet-ZnBfR, respectively, on days 3 and 5 (i.e., the diet not received on days 2 and 4). Zinc stable isotope tracer techniques will be used to measure the fractional absorption of zinc, in which tracer : tracee ratios will be measured in spot urine samples following administration of an intravenously administered tracer (68Zn) and one of two oral tracers (70Zn, 67Zn) provided with test meals over a four-day period.

Outcome measures/variables: Intake of total dietary zinc (TDZ) and phytate for each subject will be calculated during the clinical study. Fractional absorption of zinc (FAZ) will be determined from the isotopic ratios obtained in urine samples using the following equation, which shows, as an example, the calculation that will be used for zinc absorption from the diet traced with 67Zn:

FAZ = 67Zn tracer:tracee ratio / 68Zn tracer:tracee ratio * (68Zn dose given IV / 67Zn dose given orally)

Total absorbed zinc (TAZ) for each child will be calculated as follows:

TAZ (mg/d) = TDZ (mg/d) * FAZ

ELIGIBILITY:
Inclusion Criteria:

Weight for Height Z-Score (WHZ) and Height for Age (HAZ): >-2 Z-Score

No longer breastfed

No H/O diarrhoea in last 14 days

Given anti-helminthics in last three months

Exclusion Criteria:

Not meeting the inclusion criteria.

Ages: 36 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Total absorbed zinc | 13 days
  Total absorbed zinc (TAZ) for each child will be calculated as follows:
  TAZ (mg/d) = Total Dietray Zinc (TDZ) (mg/d) * Frcational Absorbed Zinc (FAZ)

CONTACTS AND LOCATIONS:
Locations (1):
- International Centre for Diarrhoeal Disease Research , Bangladesh (icddr,b), Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided